CLINICAL TRIAL: NCT03662282
Title: Omegaven as Alternative Parenteral Fat Nutrition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00033519
Record Dates: First submitted 2018-07-23; First posted 2018-09-07 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2019-07

CONDITIONS: Cholestasis; Cholestasis of Parenteral Nutrition
Keywords: Omegaven; parenteral nutrition; Liver disease; Cholestasis
MeSH Terms: conditions — Cholestasis; Hyperphagia; Liver Diseases | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug - Omegaven® (Experimental): Therapy with Omegaven® will be initiated at the goal dose of 0.5-1/kg/day. The default is over 24 hours, but shorter intervals may be considered if a program of total parenteral nutrition cycling is recommended. Omegaven® will be infused intravenously through either a central or peripheral catheter.
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Omegaven® fat emulsion will be used as a compassionate use treatment for critically ill infants with parenteral nutrition associated liver injury

SUMMARY:
To provide Omegaven® as a compassionate treatment for critically ill infants with parenteral nutrition associated cholestasis

DETAILED DESCRIPTION:
An intermediate population, Investigational New Drug study, to provide an alternate intravenous fat nutrition, Omegaven®, to help improve liver function while providing adequate nutrition for critically ill infants with parenteral nutrition associated cholestasis

ELIGIBILITY:
Inclusion Criteria:

* Greater than 14 days old
* Has parenteral nutrition associated cholestasis defined as at least 2 consecutive direct bilirubin >2 mg/dL with anatomical or functional short gut (OR >4 mg/dL if intact intestine) obtained at least 1 week apart with a ratio of direct: total bilirubin > 0.4
* Patient is parenteral nutrition dependent (unable to meet nutritional needs solely by enteral nutrition) and are expected to require parenteral nutrition for at least 3 more weeks
* Patient has not responded to other therapeutic approaches for parenteral nutrition-associated liver disease such as : cycling of parenteral nutrition, avoiding overfeeding, reduction/removal of copper and manganese from parenteral nutrition, advancement of enteral feeding, and use of Ursodiol
* Patient has been on at least 2 weeks of SMOFLIPIDs with no improvement or worsening of direct bilirubin levels
* Signed patient informed consent
* The patient is expected to have a reasonable possibility of survival
* No other known etiology of cholestasis other than parenteral nutrition-associated liver disease at the time of Omegaven® initiation

Exclusion Criteria:

* Known causes of cholestasis other than parenteral nutrition-associated liver disease including but not limited to Hepatitis C, Cystic fibrosis, biliary atresia, and alpha 1 antitrypsin deficiency are present, prior to Omegaven® initiation
* Known fish or egg allergy
* Any of the contraindications to use of Omegaven®:

  1. Active new infection at the time of initiation of Omegaven®
  2. Hemodynamic instability
  3. Recent use of medications with associated risk of bleeding, including NSAIDs
  4. Active coagulopathy or bleeding
  5. Platelet counts persistently under 30,000 despite transfusions
  6. Unstable hyperglycemia
  7. Impaired lipid metabolism (triglycerides >1000 mg/dL) while on 1 g/kg/day or less of Intralipid
  8. History of severe hemorrhagic disorders (ie. hemophilia, Von Willebrand disease, etc.)
  9. Unstable diabetes mellitus
  10. Collapse and shock
  11. Stroke/ Embolism
  12. Cardiac infarction within the last 3 months
  13. Undefined coma status

Min Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thao Ho, DO, Principal Investigator — University of South Florida
Locations (1):
- USF Health, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants were recruited from a single NICU for compassionate use of Omegaven for cholestasis.
Pre-assignment Details: Infants were screened based on inclusion and exclusion criteria. When there was a potential candidate, an IND application is submitted to FDA.
Groups:
- Drug - Omegaven®: Participants were screened based on inclusion and exclusion criteria. If and when a participant was qualified for Omegaven treatment, we sent FDA and application for IND approval. After the approval, the participant received Omegaven daily per protocol until cholestatsis resolved.
Period: Overall Study
Arm/Group | Drug - Omegaven®
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Drug - Omegaven®: These infants were more than one month old with history of long-term TPN dependence due to intestinal problem.
Arm/Group | Drug - Omegaven®
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: days] | 45 [30 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Decrease in Direct Bilirubin Level
Description: Number of participant with decrease in direct bilirubin levels within 30 days of treatment
Time Frame: First month of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Drug - Omegaven®: Omegaven treatment group
Arm/Group | Drug - Omegaven®
Number analyzed (Participants) | 2
Participants
  decrease in bilirubin level | 2
  increase or no change in bilirubin level | 0

2. Secondary Outcome: Number of Participant With Resolution of Direct Hyperbilirubinemia
Description: Number of participant with Direct bilirubin level of <2mg/dL at discontinuation of treatment
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - Omegaven®
Number analyzed (Participants) | 2
Participants
  bilirubin <2mg/dL at discontinuing of Omegaven | 1
  bilirubin >2mg/dL at discontinuing of Omegaven | 1

3. Secondary Outcome: Number of Participant With Preservation of Length
Description: Monitoring of weekly length while the patient is receiving Omegaven® treatment
Time Frame: Weekly measurement during treatment. Evaluation every 30 days from treatment initiation until discontinuation of treatment, patient hospital discharge, whichever comes first, or up to 6 months following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - Omegaven®
Number analyzed (Participants) | 2
Participants
  Preservation of length growth | 2
  fail in length growth | 0

4. Secondary Outcome: Number of Participant With Preservation of Head Circumference
Description: Monitoring of weekly head circumference while the patient is receiving Omegaven® treatment
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - Omegaven®
Number analyzed (Participants) | 2
Participants
  preservation of head circumference | 2
  Fail in head circumference growth | 0

5. Secondary Outcome: Number of Participant With Preservation of Normal Weight Gain
Description: Monitoring of daily weight gain while the patient is on Omegaven®
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - Omegaven®
Number analyzed (Participants) | 2
Participants
  preservation of weight gain | 2
  fail in weight gain | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Drug - Omegaven®
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03662282/Prot_001.pdf